CLINICAL TRIAL: NCT07025226
Title: MC230715 Pilot Study of the Mechanistic Feedback From CNS Tumors With Latent Residual Disease to Guide Individualized Therapies
Brief Title: Sequential Treatments or Combinations Including Dasatinib, Quercetin, Fisetin and/or Temozolomide for the Treatment of Previously Treated Glioma With Residual Disease
Acronym: Senolytics
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC230715; NCI-2025-03841 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-008241 (Other: Mayo Clinic Institutional Review Board); MC230715 (Other: Mayo Clinic)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Specimen Handling; Dasatinib; fisetin; fluorodopa F 18; Magnetic Resonance Spectroscopy; Watchful Waiting; Observation; Quercetin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Regimen 1 (rest, no treatment) (Active Comparator): Patients receive rest and take no treatment on days 1-35 of cycle 1. Patients at the end of cycle 1 proceed to regimen 2. Additionally, patients undergo MRI throughout the study as well as undergo blood and CSF sample collection on study. Patients may undergo 18F-DOPA-PET scans on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Other: Patient Observation; Procedure: Positron Emission Tomography
- Regimen 2 (dasatinib, quercetin) (Experimental): Patients receive dasatinib PO QD on days 1-2 and quercetin PO QD on days 1-2 of each cycle. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients without a PR or CR on imaging at the end of cycle 1 proceed to regimen 3. Patients with a PR or CR may remain on the current regimen. Additionally, patients undergo MRI throughout the study as well as undergo blood and CSF sample collection on study. Patients may undergo 18F-DOPA-PET scans on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Dasatinib; Drug: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Quercetin
- Regimen 3 (fisetin) (Experimental): Patients receive fisetin PO QD on days 1-2 of each cycle. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients without a PR or CR on imaging at the end of cycle 1 proceed to regimen 4. Patients with a PR or CR may remain on the current regimen. Additionally, patients undergo MRI throughout the study as well as undergo blood and CSF sample collection on study. Patients may undergo 18F-DOPA-PET scans on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Fisetin; Drug: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography
- Regimen 4 (temozolomide) (Experimental): Patients receive temozolomide PO QD on days 1-5 of each cycle. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients without a PR or CR on imaging at the end of cycle 1 proceed to regimen 5. Patients with a PR or CR may remain on the current regimen. Additionally, patients undergo MRI throughout the study as well as undergo blood and CSF sample collection on study. Patients may undergo 18F-DOPA-PET scans on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Temozolomide
- Regimen 5 (dasatinib, quercetin, temozolomide) (Experimental): Patients receive temozolomide PO QD on days 1-5, quercetin PO QD days 14-15 and dasatinib PO QD on days 14-15 of each cycle. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients without a PR or CR on imaging at the end of cycle 1 proceed to regimen 6. Patients with a PR or CR may remain on the current regimen. Additionally, patients undergo MRI throughout the study as well as undergo blood and CSF sample collection on study. Patients may undergo 18F-DOPA-PET scans on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Dasatinib; Drug: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Quercetin; Drug: Temozolomide
- Regimen 6 (fisetin, temozolomide) (Experimental): Patients receive temozolomide PO QD on days 1-5 and fisetin PO QD on days 14-15 of each cycle. Cycles repeat every 35 days in the absence of disease progression or unacceptable toxicity. Patients without a PR or CR on imaging at the end of cycle 1 proceed to end of study treatment and study follow up. Patients with a PR or CR may remain on the current regimen. Additionally, patients undergo MRI throughout the study as well as undergo blood and CSF sample collection on study. Patients may undergo 18F-DOPA-PET scans on study.
  Interventions: Procedure: Biospecimen Collection; Drug: Fisetin; Drug: Fluorodopa F 18; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Drug: Temozolomide

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and CSF sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Dasatinib — Given PO
  Other Names: BMS 354825; BMS-354825; BMS354825; Dasatinib Hydrate; Dasatinib Monohydrate; Sprycel
  Arms: Regimen 2 (dasatinib, quercetin); Regimen 5 (dasatinib, quercetin, temozolomide)
Drug: Fisetin — Given PO
  Other Names: 3,3',4',7-Tetrahydroxyflavone; 7,3',4'-Flavon-3-ol
  Arms: Regimen 3 (fisetin); Regimen 6 (fisetin, temozolomide)
Drug: Fluorodopa F 18 — Undergo 18F-DOPA-PET scan
  Other Names: (18F)FDOPA; 18F-DOPA; 18F-FDOPA; 3-(2-Fluoro-(sup 18)F-4,5-dihydroxyphenyl)-L-alanine; 6-(18F)Fluoro-L-DOPA; Fluorine F 18 Fluorodopa; Fluorine-18-fluoro-L-DOPA; Fluorodopa (18F); FLUORODOPA F-18; L-6-(18F)Fluoro-DOPA
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Other: Patient Observation — Receive rest and take no treatment
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Regimen 1 (rest, no treatment)
Procedure: Positron Emission Tomography — Undergo 18F-DOPA-PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Drug: Quercetin — Given PO
  Other Names: 2-(3,4-dihydroxyphenyl)-3,5,7-trihydroxy-4H-1-benzopyran-4-one; 2-(3,4-dihydroxyphenyl)-3,5,7-trihydroxy-chromen-4-one; C.I. Natural Yellow 10
  Arms: Regimen 2 (dasatinib, quercetin); Regimen 5 (dasatinib, quercetin, temozolomide)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Gliotem; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temizole; Temodal; Temodar; Temomedac; TMZ
  Arms: Regimen 4 (temozolomide); Regimen 5 (dasatinib, quercetin, temozolomide); Regimen 6 (fisetin, temozolomide)

SUMMARY:
This early phase I trial tests the safety, side effects and how well medication combinations of dasatinib, quercetin, fisetin and temozolomide work in treating patients with glioma for which the patient has received treatment in the past (previously treated) and for tumor cells that remain after attempts to treat the tumor have been made (residual disease). Dasatinib is in a class of medications called tyrosine kinase inhibitors. It works by blocking the action of an abnormal protein that signals tumor cells to multiply, which may help keep tumor cells from growing. Quercetin and fisetin are compounds found in plants. They have antioxidant and anti-inflammatory properties and help remove senescent cells, older or damaged cells that have stopped dividing but don't die off as they should and build up in tissues over time. Senescent cells may cause inflammation or damage to nearby healthy cells. Temozolomide is in a class of medications called alkylating agents. It works by damaging the cell's deoxyribonucleic acid (DNA) and may kill tumor cells and slow down or stop tumor growth. Giving medication combinations of dasatinib, quercetin, fisetin and temozolomide may be safe, tolerable and/or effective in treating patients with previously treated glioma with residual disease.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Prior diagnosis of a glioma treated with chemotherapy and/or radiation with stable disease based on Response Assessment in Neuro-Oncology (RANO) criteria

  * Must have IDH-mutant OR MGMT-methylated glioma

    * NOTE: Patients with any radiographic evidence of residual disease are eligible
* Eastern Cooperative Oncology Group (ECOG) of 0, 1, or 2, and Karnofsky performance status >= 50
* Hemoglobin ≥ 9.0 g/dL (≤ 15 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (≤ 15 days prior to registration)
* Platelet count ≥ 100,000/mm^3 (without transfusion ≤ 7 days preceding lab assessment) (≤ 15 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 2.5 x upper limit of normal (ULN) (or ≤ 5 x ULN for patients with liver involvement) (≤ 15 days prior to registration)
* Calculated creatinine clearance ≥ 45 ml/min using the Cockcroft-Gault formula (≤ 15 days prior to registration)
* Average corrected QT interval (QTc) ≤ 450 ms on triplicate 12 lead electrocardiogram (ECG) ≤ 29 days prior to registration

  * NOTE: QTc intervals will be corrected using Fridericia's formula (Fridericia 1920)
* Negative serum pregnancy test is required for persons of childbearing potential ≤ 8 days prior to registration
* Presence of an implanted cranial CSF access device, such as Ommaya reservoir or ventriculoperitoneal shunt
* Willingness to provide blood and CSF samples for research
* Co-enrollment on the neuro-oncology biorepository [institutional review board (IRB) 12-003458] for collection of research blood and CSF samples
* Provide written informed consent
* Willingness to return to Mayo Clinic for follow-up

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential and persons able to father a child who are unwilling to employ adequate contraception
* Patients who are not appropriate medical candidates due to current or past medical history or uncontrolled concurrent illness which limits safety of or compliance to study proceedings
* Participants who are unable to swallow tablets or who are at risk for impaired absorption of oral medication

  * NOTE: This includes but not limited to, refractory vomiting, gastric resection/bypass, or duodenal/jejunal resection
* Patients with known hypersensitivity or allergy to all of the study drugs on the protocol (known hypersensitivity or allergy to one drug does not preclude participation in this protocol)
* Inability to undergo MRI scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Completion of 3 cycles | Up to 16 weeks
  Will evaluate feasibility of serially screening multiple candidate therapies or combinations based on individualized empiric biological feedback from biospecimens and imaging. This will be measured as the percentage of patients successfully completing 3 cycles of drug administration (study visits). A cycle is 35 +/- 7 days. Regimen will be considered feasible if at least 2/3 of patients can achieve this target.
Turnaround time for scan and marker data | Up to 16 weeks (completion of 3 cycles)
  Will also evaluate feasibility as the turnaround time for scan and marker data that is used to determine if patients should stay on current therapy or move to the next regimen. The outcomes will be cycle-specific. A cycle is 35 +/- 7 days. The target for this is a mean turnaround time of 3 days; if the maximum turnaround time exceeds 5 days, this will prompt an evaluation of process to identify barriers.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 3 years
  Will assess the safety of this algorithm-based approach to individualized therapeutic drug combinations in patients with pre-recurrent central nervous system tumors. The study drugs will be considered well-tolerated with no grade 3 or higher adverse event attributable to the drugs in the 10 patients. Adverse events will be evaluated per the Common Terminology Criteria for Adverse Events (CTCAE) version 5 criteria and summarized by type and severity as well as perceived attribution to study treatment for each of the regimens received by patients.
Change in senescence-associated proteins | Baseline; up to 3 years
  Will evaluate relative change from baseline in enrichment for a panel of senescence-associated proteins in cerebrospinal fluid (CSF) for each sequentially administered senolytic agent. An effective senolytics regimen will decrease CSF senescence associated secretory phenotype, including monocyte chemoattractant protein-1 levels, by at least 25%.
Cell-free mitochondrial deoxyribonucleic acid (DNA) | Baseline; up to 3 years
  Will evaluate the percentage change in cell-free mitochondrial DNA. An effective senolytics regimen will decrease cell-free mitochondrial DNA by at least 25%.
2-Hydroxyglutarate (2-HG) | Baseline; up to 3 years
  Will evaluate the percentage change in 2-HG.
Amplified DNA junctions | Baseline; up to 3 years
  Will evaluate the percentage change in amplified DNA junctions (if applicable).
Volume of disease | Baseline; up to 3 years
  Will evaluate the percentage change in the volume of disease above a tumor to normal standardized uptake value maximum ratio of 2 from fluorodopa F 18-positron emission tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Terence C. Burns, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials
- See also: Review article discussing the rationale for and general design of this study — https://pubmed.ncbi.nlm.nih.gov/38030881/